CLINICAL TRIAL: NCT04381390
Title: Comparison of Whole Eggs vs. Egg Whites Consumption on Regulatory Myokines, Muscular Strength, Hypertrophy, Power and Body Composition.
Brief Title: Egg Consumption and Muscular Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexei Wong (Other)
Collaborators: Tehran University (Unknown)
Responsible Party: Sponsor-Investigator, Alexei Wong, Assistant Professor, Marymount University
Organization: Marymount University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 11/27498
Record Dates: First submitted 2020-05-01; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Hypertrophy
MeSH Terms: conditions — Hypertrophy | interventions — Resistance Training; Egg White

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole egg consumption (Experimental): This arm involved whole egg consumption concomitant with 12 weeks of resistance training. Subject ingested three whole eggs per day immediately after resistance training.
  Interventions: Dietary Supplement: Whole egg and resistance training
- Egg whites consumption (Experimental): This arm involved egg white consumption concomitant with 12 weeks of resistance training. Subject ingested an isonitrogenous quantity of six egg whites per day immediately after resistance training.
  Interventions: Dietary Supplement: Egg whites and resistance training

INTERVENTIONS:
Dietary Supplement: Whole egg and resistance training — This intervention consisted of whole egg consumption concomitant with 12 weeks of resistance training. Subject ingested three whole eggs per day immediately after resistance training.
  Arms: Whole egg consumption
Dietary Supplement: Egg whites and resistance training — This intervention consisted of egg white consumption concomitant with 12 weeks of resistance training. Subject ingested an isonitrogenous quantity of six egg whites per day immediately after resistance training.
  Arms: Egg whites consumption

SUMMARY:
Eggs may be a viable alternative to various types of supplemental proteins given its similar ratings on various measures of dietary protein quality.

The investigators hypothesis is that whole eggs would create a greater improvement in skeletal regulatory markers, hormonal responses and body composition than egg white ingestion in resistance-trained men.

DETAILED DESCRIPTION:
The aim of this investigation was to compare the effects of whole egg versus egg white ingestion (daily and after training sessions) during 12 weeks of resistance training on skeletal muscle regulatory markers, hormonal responses and body composition in resistance-trained men. Specific aims of the study are to:

To investigate the extent to which both whole egg and egg white ingestion will improve anabolic factors, fat free mass, fat mass and decrease catabolic markers after 12 weeks of resistance training in resistance-trained men.

ELIGIBILITY:
Inclusion Criteria:

* performing resistance training at least three times a week for 1 year prior to the start of the study
* not taking any dietary supplements or medications for at least 1 year prior to the start of the study
* no known medical issues
* no alcohol consumption or smoking for at least 1 year prior to the start of the study
* no egg allergy/sensitivity.

Exclusion Criteria:

* non-willingness to continue nutritional or exercise protocols
* participation in exercise other than the prescribed resistance training program
* consumption of dietary supplement (other than egg) during the study period
* Missing more than one resistance training session or post-exercise egg consumption throughout the study period

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Circulatory Myokines levels | 12 weeks
  Fasting blood samples were collected from the antecubital vein using standard procedures and then analized to establish concentration of myostatin, follistatin, FGF-2, TGF-β1 and ACVA.
Circulatory hormone levels | 12 weeks
  Fasting blood samples were collected from the antecubital vein using standard procedures and then analized to establish concentrations of testosterone, IGF-1, insulin and cortisol
Muscle mass | 12 weeks
  Skeletal muscle mass will be evaluated using computed tomography
Body fatness | 12 weeks
  Body fat will be evaluated using bioelectrical impedance

SECONDARY OUTCOMES:
Muscular Strength | 12 weeks
  Using 1 repetition maximum

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Wong, Principal Investigator — Marymount University
Locations (1):
- Marymount University, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bagheri R, Hooshmand Moghadam B, Ashtary-Larky D, Forbes SC, Candow DG, Galpin AJ, Eskandari M, Kreider RB, Wong A. Whole Egg Vs. Egg White Ingestion During 12 weeks of Resistance Training in Trained Young Males: A Randomized Controlled Trial. J Strength Cond Res. 2021 Feb 1;35(2):411-419. doi: 10.1519/JSC.0000000000003922. PMID 33306586